CLINICAL TRIAL: NCT00494403
Title: Effects of Ankle Instability on Cervical Proprioception
Brief Title: Chronic Ankle Instability and Proprioception
Status: Completed | Type: Observational
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Principal Investigator, Dennis Enix, DC, MBA, Assistant Professor, Logan College of Chiropractic
Other Study IDs: RD0615070095; 6
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Ankle Sprains
Keywords: sprain proprioception

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this investigation is to determine the effects of chronic ankle instability on cervical spine and knee proprioception as measured using joint position sense to investigate whether correlation can be drawn between the two.

ELIGIBILITY:
Inclusion Criteria:

* History of ankle instability
* Ages 20-65 yoa Exclusion Criteria: - Recent surgery, have any unstable or fused joints of the cervical spine.
* Medications, prescription or herbal muscle stimulants, relaxants.
* Any previ

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort of college aged students with a history of ankle sprains.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
joint repositioning error | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Logan University, College of Chiropractic, St Louis, Missouri, United States